CLINICAL TRIAL: NCT01569035
Title: a Randomized Clinical Trial Using Oral Anti Coagulant in the Management of Unexplained Oligohydramnios
Brief Title: Warfarine in Unexplained Oligohydramnios
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, doctor, Woman's Health University Hospital, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: wuoh
Record Dates: First submitted 2012-03-24; First posted 2012-04-02 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Oligohydramnios
Keywords: oligohudramnios; oral anti coagulant; Dopplar ultrasound
MeSH Terms: conditions — Oligohydramnios | interventions — Warfarin; Coumarins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- warfarin (Active Comparator): oral anti coagulant
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin — 3 mg warfarin oral tablet for 2 to 3 weeks
  Other Names: coumarins

SUMMARY:
This study examines using oral anti coagulant warfarin in the management of unexplained oligohydramnios improve the perinatal outcome with little or no complications to the mother or the neonates.

DETAILED DESCRIPTION:
A randomized controlled study with 200 pregnant women with idiopathic oligohydramnios between 28 and 32 weeks. Women were randomized to receive 3 mg warfarin daily (Warfarin group) or placebo (Placebo group). Outcomes included amniotic fluid index (AFI), duration of pregnancy and perinatal outcomes including Apgar score, Neonatal intensive care admission (NICU).

Patients were eligible for inclusion if they were 28t to 32 weeks of pregnancy and age 18-35 years and diagnosed to have idiopathic oligohydramnios excluded by medical history and detailed u/s examination,the cut off AFI was less than 5cm. A written informed consent was taken. Gestational age was determined on the basis of the last menstrual period, confirmed by an ultrasound scan conducted between 6 and 14 weeks of gestation The clinical work-up included a history taken prior to enrollment, examination, obstetric ultrasound evaluation, and biophysical profile taken after 32 weeks of pregnancy Exclusion criteria were chronichypertension, anaemia ,cardiac diseases ,or history of premature rupture of membrane or structural malformations. Sterile speculum examination was done to exclude rupture of membrane. Detailed level 2D ultrasonography to determine the possible etiology and to exclude the multiple pregnancy and fetal death. All fetuses were alive with fetal weight were prior treatment and each follow up visits. Doppler ultrasound for uterine, umbilical and middle cerebral arteries, and fetal ascending aorta was done using resistant index (RI), pulsetilty index (PI) and systolic/diastolic (S/D) ratio before and in each follow up visits. Laboratory tests were obtained included complete blood picture, liver function test, immunological tests to exclude antiphospholipid antibodies was done. After these all patients with unknown major cause were classified as idiopathic oligohydramnios and the treatment started to them.

The patients were randomly allocated to 2 treatment groups using computer-generated numbers in sealed envelopes. Treatment was started immediately after the test result was known, and continued until 36 completed weeks of pregnancy or active onset of labor. The patients were randomized to receive either a daily dose of 3 mg warfarin oral tablet or a daily placebo sachet The placebo sachets were especially manufactured to look identical to warfarin tablets. The tablets were placed in sacs and then stored in envelopes numbered from 1 to 200 The envelopes were numbered and randomized according to computer-generated randomization tables to ensure an equal number of patients in each arm. Throughout the trial, access to the randomization code was available only to the pharmacist who manufactured the placebo and packed the envelopes and was not available to any of the treating physicians or patients

Treatment protocol:

One tablet of 3 mg of warfarin was provided daily to each patient in Warfarin group and placebo to Placebo group. After starting the treatment; weekly follow up of the patient for four weeks till 36 weeks and 2 weeks thereafter. Each follow up visit the following were done; assessment of the amniotic fluid, biophysical profile including non stress test (NST), Doppler U/S of fetal ascending aorta, uterine, middle cerebral and umbilical arteries. Laboratory measurement of prothrombine time and concentration and INR are checked daily until in the therapeutic range for 2 consecutive days, then twice a week for 1-2 weeks, then weekly until stable. Change in a patient's condition, e.g. liver disease, intercurrent illness, and new drug started necessitates more frequent testing. Patients should be advised to report any bruising or bleeding immediately, as advised, avoid aspirin but use paracetamol for pain ,avoid contact sports and activities carrying a risk of head injury. During labor or cesarean section visual inspection of blood loss and 48 hours follow up for the occurrence of hematomas and neonatal follow up for any bleeding problems. Discontinuation of treatment was done if after two weeks of treatment no changes of the amniotic fluid, manifestation of fetal distress appeared or the patient completed 36 weeks of gestation.

Assessment of outcome measures The primary outcome was improvement of the amniotic fluid and improving the biophysical profile. The secondary outcome is prolongation of pregnancy till suitable time of fetal maturity. The baseline characteristics of the study participants were analyzed including amniotic fluid index, Doppler indices changes of the fetal and maternal vessles, mode of the delivery and the rate of continuation of pregnancy. Finally, the maternal and neonatal complications and the cost of the treatment were calculated.

Statistical analysis:

. Data collected and analyzed by computer program SPSS version 17 Chicago -USA

* Data expressed as mean ± S.D, number and percentage
* Using Paried t.test to determine significance for numeric variable
* Using Pearson´s correlation to determine significance between variables N.S= P > 0.05 No significance

  * = P < 0.05 Significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were 28th to 32nd weeks of pregnancy and
* age 18-35 years and
* diagnosed to have idiopathic oligohydramnios excluded by medical history and
* detailed u/s examination,
* the cut off AFI was less than 5cm

Exclusion Criteria:

* Exclusion criteria were chronic hypertension,
* anaemia,
* cardiac diseases,or
* history of premature rupture of membrane or
* structural malformations.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome was improvement of the amniotic fluid and improving the biophysical profile | 2 to 3 three weeks
  The primary outcome was improvement of the amniotic fluid and improving the biophysical profile

SECONDARY OUTCOMES:
The secondary outcome is prolongation of pregnancy till suitable time of fetal maturity | 4 weeks
  The baseline characteristics of the study participants were analyzed including amniotic fluid index, Doppler indices changes of the fetal and maternal vessles, mode of the delivery and the rate of continuation of pregnancy. Finally, the maternal and neonatalcomplications and the cost of the treatment were calculated.intention to treat analysis is done.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M.D, Principal Investigator — Women Health Hospital
Locations (1):
- Women Health Hospital, Asyut, Egypt